CLINICAL TRIAL: NCT06193161
Title: Feasibility and Preliminary Efficacy of Internet Delivered Prolonged Exposure Immigrants With PTSD: a Randomized Controlled Trial
Brief Title: Prolonged Exposure for Swedish Immigrants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Bragesjo, Principal investigator, Clinical psychologist, PhD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-02715-01
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; digital treatment; therapist-guided treatment; migrants; prolonged exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are randomized to I-PE for eight weeks or to a waitlist. Participants in the control arm will be crossed over to I-PE treatment after completion of the 1 month follow up (primary endpoint).
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapist-guided internet delivered prolonged exposure (Experimental): Therapist-supported internet delivered prolonged exposure comprising psychoeducation about PTSD, controlled breathing, imaginal exposure including processing, in vivo exposure and relapse prevention. The treatment will be delivered in a digital platform for eight weeks. Participants will have access to a therapist that will guide them through treatment in a text based format.
  Interventions: Behavioral: Therapist-supported internet delivered prolonged exposure
- Waiting list (No Intervention): Waiting list up for eight weeks and up until the 1-month follow up.

INTERVENTIONS:
Behavioral: Therapist-supported internet delivered prolonged exposure — Therapist-supported internet delivered prolonged exposure for eight weeks.
  Arms: Therapist-guided internet delivered prolonged exposure

SUMMARY:
The goal of this clinical trial is to compare therapist-guided internet delivered prolonged exposure (I-PE) in simple english to a waiting list condition for immigrants in Sweden diagnosed with post-traumatic stress disorder (PTSD).

The main objectives are to establish feasibility and preliminary efficacy of I-PE for immigrants with PTSD in a single-blind, parallel-group superiority Randomized Controlled Trial (N=100) comparing I-PE with a waiting-list condition, starting with a nested pilot (N=30) to ensure feasible and acceptable recruitment and treatment strategies. Study participants will be randomly assigned to either eight weeks of I-PE or a waiting-list for the same amount of time on a 1:1 ratio without restriction. Feasibility and acceptability data will be reported including recruitment rate, sample demographics, data attrition, treatment adherence and a detailed dropout analysis. A preliminary investigation of the within-group effect size will also be conducted. Recruitment is designed to be broadly inclusive with minimal exclusion criteria.

DETAILED DESCRIPTION:
There is an urgent need for dissemination of evidence-based treatments for PTSD beyond the Swedish language criteria and developed in an easy-to-read manner and develop the treatment so that it can be easily made available to a large number of afflicted who are excluded from treatment.The overall aim of the study is to evaluate I-PE for immigrants with PTSD living in Sweden who can read and write easy English. The treatment will be written in easy English and adapted to the target population with regards to specific contextual characteristics.

The study is a single-blind, parallel-group superiority randomized controlled trial with 100 participants that will compare I-PE with a waiting list condition. The primary outcome is the self-rated Posttraumatic Stress Disorder Checklist version 5 (PCL-5) at the 1-month follow up. Secondary outcomes are the blind-rater administered Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), self-rated symptoms of depression quality of life, dropout rate, level of health care utilization, satisfaction with treatment and negative effects. Patients in the control arm will be crossed over to I-PE treatment after completion of the 1 month follow up (primary endpoint). Assessments will be conducted pre-treatment, post-treatment, 1 month (primary endpoint) and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of PTSD, according to the diagnostic criteria based on Diagnostic and statistical manual of mental disorders, 5th edition (DSM-5; American Psychiatric Association, 2013)
* ≥ 18 years
* Able to read and write in English
* Immigrant residing in Sweden
* Able to provide digital informed consent
* Daily access to a computer or device with internet connection

Exclusion Criteria:

* PTSD is not the primary treatment concern
* Initiation or adjustment of any psychotropic medication within the last 4 weeks prior to commencement of treatment
* Serious mental health symptoms, such as mania, psychosis, alcohol, or substance use disorders or current suicide risk warranting immediate clinical attention.
* Ongoing trauma-focused CBT or Eye movement desensitization and reprocessing therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, through the treatment period up to eight weeks, and 1-month and 6-month after treatment completion.
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS-5) | Baseline up to 1-month after treatment completion
  The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in depression as assessed by The Patient Health Questionnaire (PHQ-9) | Baseline, immediately after treatment completion, 1-month and 6-month after treatment completion
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in general quality of life assessed by 12-Item Short-Form Health Survey (SF-12) | Baseline, immediately after treatment completion, 1-month and 6-month after treatment completion
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Scores range from 0 to 100. A higher score means higher health.
Treatment credibility assessed by the Credibility/expectancy scale (CEQ) | Treatment week 3 (three weeks from baseline).
  Measures treatment expectancy and rationale credibility. The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Change in stigma and barriers related to mental health and competency in mental health assessed by the Stigma-9 Questionnaire (STIG-9), | Baseline, immediately after treatment completion and 1-month after treatment completion
  The STIG-9 consists of nine items assessing cognitive, behavioural and affective aspects of perceived mental health-related stigma. The item responses are summarized in a sum score ranged 0-27 points. Higher scores indicate stronger expectations of negative societal beliefs, feelings, and behaviours towards 'mentally ill' people.
Change in stigma and barriers related to mental health and competency in mental health assessed Barriers to Access to Care Evaluation Scale (BACES) | Baseline, immediately after treatment completion and 1-month after treatment completion
  The Barriers to Access to Care Evaluation (BACE) is a 30-item measure scored from 0 (not at all) to 3 (a lot) with higher scores indicating a greater barrier.
Change in stigma and barriers related to mental health and competency in mental health assessed Mental Health Knowledge Schedule (MHKS) | Baseline, immediately after treatment completion and 1-month after treatment completion
  MHKS is a twelve-item scale comprising domains of relevant evidence-based knowledge in relation to stigma toward mental illness. Items are coded on an ordinal scale (1-5). Items which the respondent strongly agrees with score 5 points; 1 point reflects a response to which the respondent strongly disagrees. The total score is calculated by adding the points obtained for each of the 12 items. Higher total scores correspond to greater knowledge
Change in Treatment inventory of costs associated with psychiatric illness (TIC-P) | Baseline, immediately after treatment completion and 1-month after treatment completion
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder. The TIC-P questionnaire measures costs in two dimensions: use of health resources and loss of productivity. Lower cost is better.
Treatment satisfaction measured by the Client Satisfaction Questionnaire (CSQ-8 | Immediately after treatment completion
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Treatment satisfaction measured by the Internet Evaluation and Utility Questionnaire (IEUQ) | Immediately after treatment completion
  The Internet Evaluation and Utility Questionnaire (IEUQ) is a 13-item measure that examines the participants' experiences of a web-based intervention. Score range from 0-72. Higher values indicating higher satisfaction.
Adverse events related to treatment measured by the Negative effects questionnaire-20. | 1-mont after treatment completion
  Self-rated questionnaire on negative effects. It contains 20 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.

OTHER OUTCOMES:
Number of completed treatment modules | Baseline up to treatment completion at 8 weeks
  Data will be gathered on total number of completed modules during the 8 week treatment.
Number of messages sent and received in the digital platform | Baseline up to treatment completion at 8 weeks
  Data will be gathered on total number of messages sent and received back and forth between the participant and the therapist during the 8 week treatment.
Experience with the digital treatment as assessed by qualitative interviews | Immediately after treatment completion
  During the nested study phase a subsample of the participants (N=5-15) will be interviewed at post-treatment regarded treatment comprehension, language adaptions and relevance.
The proportion of participants that conducts the weekly measures and further assessment points | Baseline up to 6-month after treatment completion
  The proportion of participants that conducts the weekly measures and further assessment points
Number of drop-outs from treatment | Completion of the treatment period, up to 8 weeks
  Number of drop-outs from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molander O, Kolaas K, Jayaram-Lindstrom N, Ponten M, Sarnholm J, Bragesjo M. Mind the gap: a nested randomised pilot study of culturally inclusive, internet-delivered prolonged exposure for PTSD among immigrants. Eur J Psychotraumatol. 2025 Dec;16(1):2520637. doi: 10.1080/20008066.2025.2520637. Epub 2025 Jun 30. PMID 40587567